CLINICAL TRIAL: NCT02681744
Title: Effects of Resistance Training on Sarcopenic Obesity Index in Older Women: a RCT.
Brief Title: Sarcopenia, Obesity, and Resistance Training
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Brasilia (Other)
Responsible Party: Principal Investigator, Ricardo Moreno Lima, PhD, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 487622/2012-0
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-02

CONDITIONS: Sarcopenia; Aging; Obesity
MeSH Terms: conditions — Sarcopenia; Obesity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (No Intervention): These participants will be instructed to maintain their habits during 24 weeks. Before and after the aforementioned period, they will be asked to perform body composition and strength assessments, using DXA and isokinetic dynamometer, respectively.
- Experimental group (Experimental): Participants from the experimental group will assign to the resistance training program undergo physician screening at rest and under cardiopulmonary exercise test conditions before starting the program. Following a three-week familiarization process, participants undergo one repetition maximum (1-RM) testing for each of the exercises of the training program. This procedure intended to determine exercise load and will be systematically repeated in four-week intervals. Volunteers will train thrice per week during 24 weeks. The training program will involve the following exercises: chest press, lat pulldown, knee extension, hamstrings curl, leg press, hip abduction.
  Interventions: Behavioral: Resistance Training

INTERVENTIONS:
Behavioral: Resistance Training — 24-weeks of progressive strength training
  Other Names: Strength Training
  Arms: Experimental group

SUMMARY:
The purpose of this study was to examine the effects of resistance training on sarcopenic obesity in older women.

DETAILED DESCRIPTION:
To examine the effects of resistance training on sarcopenic obesity in older women, a representative sample of older women from Brasília, Brazil (n>244 subjects), will be recruited and invited to undergo body composition measurement using dual-energy x-ray absorptiometry. Moreover, the Sarcopenic Obesity index and isokinetic strength evaluations will be performed. It will be a single-blind randomized, controlled 24-week clinical trial, in which experimental group will receive a progressive resistance training program, meanwhile control group will receive instructions to maintain their lifestyle habits. Randomization will be conducted by computer-generated list in blocks of 10. Additionally, body composition, strength assessment, and sarcopenic index will collected and compared after the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* Community older women (aged between 60 and 80 years).

Exclusion Criteria:

* individuals with any metallic implant or artificial pacemaker, who had undergone hip surgery, who were unable to walk without assistance and those affected by metabolic or endocrine disorders that affect the muscular system.

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 244 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Laboratorial Body Composition assessment (DXA) | 30 minutes
  DXA-derived body fat and DXA-derived fat free mass

SECONDARY OUTCOMES:
Isokinetic peak torque of leg extension (dynamometer isokinetic) | 20 minutes
  Dominant leg extension peak torque will be recorded in three sets of maximal effort

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo M Lima, PhD, Principal Investigator — University of Brasilia
Locations (1):
- Faculdade de Educação Física, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Undecided